CLINICAL TRIAL: NCT06235632
Title: Policy and Training Intervention in Responsible Marijuana Sales Practices to Reduce the Risk of Selling to Intoxicated Customers
Brief Title: Responsible Marijuana Sales Practices to Reduce the Risk of Selling to Intoxicated Customers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Pacific Institute for Research and Evaluation (Other); National Opinion Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0347; 1R01AA031591-01A1 (NIH)
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Alcoholic Intoxication; Automobile Accident; Cannabis
Keywords: randomized partial cross-over trial; Responsible Marijuana Vendor training
MeSH Terms: conditions — Alcoholic Intoxication; Marijuana Abuse | interventions — Policy

STUDY DESIGN:
Intervention Model Description: This is a pretest-posttest randomized control partial cross-over trial. A subsample of stores will be randomly assigned to receive the intervention while the rest will receive the control training. After the posttest assessment is conducted, the remaining control stores will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Policy and Training Intervention (Experimental): This intervention includes the combination of a 2-hour policy meeting held by the Oregon Liquor and Cannabis Commission to teach the current laws around selling recreational marijuana as well as access to the TrainToTend program which contains 5 modules: The Laws, ID Checking, Health Effects, Customer Service, and Rules of the Trade
  Interventions: Behavioral: Policy and Training Intervention
- Usual and Customary Policy and Training (UC-PT) (Control) Condition (Active Comparator): This is basic Responsible Marijuana Vendor training currently provided by the Oregon Liquor and Cannabis Commission and includes reading a booklet on selling recreational marijuana responsibly and passing and exam
  Interventions: Behavioral: Usual and Customary Policy and Training (UC-PT) (Control) Condition

INTERVENTIONS:
Behavioral: Policy and Training Intervention — The intervention is a combination of a policy training and access to an in-depth training program to teach marijuana vendors the skills needed to refuse intoxicated customers
  Arms: Policy and Training Intervention
Behavioral: Usual and Customary Policy and Training (UC-PT) (Control) Condition — The active control training that is already provided to marijuana vendors by the Oregon Liquor and Cannabis Commission
  Arms: Usual and Customary Policy and Training (UC-PT) (Control) Condition

SUMMARY:
The new recreational marijuana markets are contributing to polysubstance-impaired driving and other harms, especially when marijuana is used in combination with alcohol, by selling marijuana to obviously-intoxicated customers. In this study, the effectiveness of an intervention to reduce the risk of marijuana sales to obviously-intoxicated customers will be tested in the state-licensed recreational marijuana market in Oregon, one of the first states to ban such sales. The intervention will combine efforts by state regulators to increase deterrence of the state law prohibiting marijuana sales to obviously-intoxicated customers with training of store personnel to recognize signs of intoxication and refuse sales. It will also include testing the rate at which visibly intoxicated customers are refused alcohol at nearby establishments that sell alcohol either on-site or off-site

DETAILED DESCRIPTION:
The new recreational marijuana markets are contributing to morbidity and mortality due to marijuana- and polysubstance-impaired driving and other harms by selling a social intoxicant (i.e., marijuana) to already intoxicated customers. Impairment increases when marijuana is combined with alcohol, making driving particularly risky and also contributing to other injuries and violence. In recreational marijuana markets, deterrence efforts to reduce impaired driving directed at drivers face challenges due to dispute over THC levels in per se laws and lack of valid field sobriety tests. An alternative prevention approach is to decrease access to marijuana by alcohol-impaired customers. The goal of this research is to test the effectiveness of a policy and training (PT) intervention in the state-licensed recreational marijuana market in Oregon, where state law bans sales to obviously-intoxicated customers. It combines policy efforts by state regulators to increase deterrence of Oregon's law and motivate store management to comply and training of store personnel in skills to recognize intoxication and refuse sales, using a responsible marijuana vendor online training developed by the research team. The specific aims of the project are to: 1) conduct pseudo-intoxicated patron (PiP) assessments at state-licensed recreational marijuana stores (n=213) in the greater Portland metropolitan area (i.e., Clackamas, Multnomah, and Washington Counties) in Year 1; 2) implement a PT intervention in Year 2 designed to increase compliance with Oregon law prohibiting sale of recreational marijuana products to obviously-intoxicated customers with a subsample of stores (n=68), assigned at random, that intends to a) make owners/managers of recreational marijuana stores aware of Oregon's law prohibiting sales of marijuana to obviously-intoxicated customers, b) increase their risk perception and motivation to comply with this law, and c) train store personnel in skills needed to recognize signs of intoxication in customers and refuse sales; 3) compare PT intervention stores to usual and customary policy and training (UC-PT) stores (n=145) in a randomized controlled trial by posttesting state-licensed recreational marijuana stores in greater Portland with PiP assessments for refusal of sales in Year 3; and 4) estimate impact of the PT intervention on refusal to PiPs by implementing the PT intervention with the remaining stores in Portland in Year 3 in a partial cross-over design and assessing state-licensed stores in greater Portland with the PiP protocol in Year 4 and in Year 5. The research is innovative and high impact by testing one of the first interventions to prevent recreational marijuana sales to obviously-intoxicated customers in one of the first states to ban such sales to reduce the risk of poly-substance impaired driving and other harms. The design allows for reproducibility by using a partial cross-over to enhance power with both between- and within-group comparisons. The PT intervention can be a model intervention to improve compliance with regulations on recreational marijuana sales in other states that have legalized recreational marijuana, now numbering 17 U.S. states, or that are considering legalization.

ELIGIBILITY:
Inclusion Criteria:

* Recreational Marijuana Stores:

  * Located in the greater Portland, Oregon metropolitan area or Salem, Oregon metro area
  * Hold an active recreational marijuana license from the Oregon Liquor Control Commission (OLCC) as of July 1, 2022
  * A retail store that sells recreational marijuana products
  * Store is open for business
  * Have a smart phone, tablet computer, or personal computer with Internet access
  * Owner or manager consent for store to participate
* Store personnel:

  * Own or employed at a state-licensed recreational marijuana store in greater Portland, Oregon or Salem, Oregon metro area
  * Sell recreational marijuana products in a retail store
  * Aged 21 or older (by state law)
  * Able to read English
  * Have a smart phone, tablet computer, or personal computer with Internet access
  * Consent to participate
* Alcohol Establishments

  * Located in the greater Portland, Oregon or Salem metropolitan area
  * Hold an active liquor license from the Oregon Liquor Control Commission (OLCC) as of July 1, 2022
  * An establishment that sells alcohol for on-site or off-site consumption
  * Store is open for business

Exclusion Criteria:

* Recreational Marijuana Stores:

  * Have an inactive, suspended, or revoked recreational marijuana license
  * Licensed to sell only medical marijuana
* Store Personnel:

  • Cannot read English
* Alcohol Establishments • Have an inactive, suspended, or revoked liquor license

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Refusal Rate of Sales of Marijuana to Obviously-intoxicated Customers | Establishments will be evaluated by PiP assessments 4 times (including baseline) over 5 years
  The rate at which establishments refuse to sell to obviously-intoxicated customers will be obtained via a pseudo-intoxicated patron (PiP) assessment

SECONDARY OUTCOMES:
Refusal Rate of Sales of Alcohol to Obviously-intoxicated Customers | Alcohol establishments will be evaluated by PiP assessments 1 time during Year 1
  The rate at which establishments refuse to sell to obviously-intoxicated customers will be obtained via a pseudo-intoxicated patron (PiP) assessment

CONTACTS AND LOCATIONS:
Overall Officials: Gill Woodall, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (1):
- Klein Buendel, Inc., Golden, Colorado, United States